CLINICAL TRIAL: NCT04832230
Title: Study of Diagnostic Biomarkers of Acute Acoustic Trauma
Acronym: BIOTSA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Direction Centrale du Service de Santé des Armées (Other)
Responsible Party: Sponsor
Other Study IDs: 2020PBMD02; 2020-A01504-35 (Other: IDRCB)
Record Dates: First submitted 2021-04-01; First posted 2021-04-05 (Actual); Last update posted 2022-11-17 (Actual); Status verified 2022-11

CONDITIONS: Acoustic Trauma
MeSH Terms: conditions — Hearing Loss, Noise-Induced | interventions — Hearing; Noise

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy individuals: This group is composed of healthy individuals without previous noise exposure.
  Interventions: Other: Hearing test; Other: Questionnaire about previous noise exposure; Other: Otoacoustic emission measurement; Other: Electrocochleography; Other: Speech audiometry in noise; Other: Multi-frequency impedance measurement; Biological: Blood sample collection
- Acute acoustic trauma patients: This group is composed of patients suffering from acute acoustic trauma.
  Interventions: Other: Hearing test; Other: Questionnaire about previous noise exposure; Other: Otoacoustic emission measurement; Other: Electrocochleography; Other: Speech audiometry in noise; Other: Multi-frequency impedance measurement; Other: Assessment of tinnitus severity; Biological: Blood sample collection

INTERVENTIONS:
Other: Hearing test — The hearing test is composed of several examinations:
  * pure tone audiogram
  * otoscopy
  * tympanometry
  Healthy individuals: The hearing test will be performed at enrollment (Day 0). Patients: The hearing test will be performed at Day 1, Day 3, Day 7 and Day 30.
Other: Questionnaire about previous noise exposure — The participant will have to fill in a questionnaire about his/her previous noise exposure at enrollment (Day 0).
Other: Otoacoustic emission measurement — Healthy individuals: Otoacoustic emission will be measured at enrollment (Day 0).
  Patients: Otoacoustic emission will be measured at enrollment (Day 0), at Day 1, Day 3, Day 7 and Day 30.
Other: Electrocochleography — Healthy individuals: Electrocochleography will be performed at enrollment (Day 0).
  Patients: Electrocochleography will be performed at Day 30.
Other: Speech audiometry in noise — Healthy individuals: Speech audiometry in noise will performed at enrollment (Day 0).
  Patients: Speech audiometry in noise will performed at enrollment (Day 0), at Day 1, Day 3, Day 7 and Day 30.
Other: Multi-frequency impedance measurement — Healthy individuals: Multi-frequency impedance will be measured at enrollment (Day 0).
  Patients: Multi-frequency impedance will be measured at Day 30.
Other: Assessment of tinnitus severity — Tinnitus severity will be assessed using a visual analogic scale at enrollment (Day 0), at Day 1, Day 3, Day 7 and Day 30.
  Groups: Acute acoustic trauma patients
Biological: Blood sample collection — Healthy individuals: A blood sample will be collected at enrollment (Day 0). Patients: A blood sample will be collected at enrollment (Day 0), at Day 1, Day 3, Day 7 and Day 30.

SUMMARY:
Every year, more than two thousand acute acoustic trauma occur in France, equally between the military and the civilian environment.

Currently, acute acoustic trauma is a pathology with no specific validated treatment, and it is the cause of many handicapping situations. Improving the future of patients requires a better understanding of the neurophysiological mechanisms of noise-induced hearing impairment. They are multiple and pure tone audiometry, the only reference examination, does not allow to differentiate them. Moreover, in the aftermath of acute acoustic trauma, pure tone audiometry tends to improve spontaneously, but this recovery is misleading, as a number of studies in animals have shown that irreversible lesions remain.

The hypothesis of this study is that it is possible to identify new entities, specific to the type of cochlear lesions, in order to clarify the diagnosis of acute acoustic trauma. These entities will be identified by the evaluation of noise-induced hearing impairment via a combination of molecular (proteomic and genomic), physiological and behavioral data. These diagnostic details may then be used to improve prevention or therapy.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40
* Healthy individuals: without hearing pathology
* Patients: acute acoustic trauma diagnosis within 72h

Exclusion Criteria:

* History of hearing pathology
* History of severe head injury
* Ototoxic drug therapy
* Abnormal otoscopy and/or tympanometry

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population is composed of healthy individuals who have never been exposed to noise and patients suffering from acute acoustic trauma.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-06-15 (Estimated); Study Completion 2024-06-15 (Estimated)

PRIMARY OUTCOMES:
Identification of diagnostic biomarkers of hearing impairment in patients suffering from acute acoustic trauma | Through study completion, an average of 3 years
  Machine learning analyses will be performed on the whole collected data to identify diagnostic biomarkers.

CONTACTS AND LOCATIONS:
Locations (14):
- France (14):
  - 102e Antenne Médicale, Angoulême
  - 38e Antenne Médicale, Bitche
  - Hôpital d'Instruction des Armées Clermont-Tonnerre, Brest
  - Laboratoire mobile d'Audition de l'Institut de Recherche Biomédicale des Armées, Brétigny-sur-Orge
  - 171e Antenne Médicale, Caylus
  - Hôpital d'Instruction des Armées Percy, Clamart
  - 41e Antenne Médicale, Dieuze
  - 123e Antenne Médicale, Guer
  - Hôpital d'Instruction des Armées Laveran, Marseille
  - 13e Antenne Médicale, Montlhéry
  - 109e Antenne Médicale, Saint-Maixent-l'École
  - 43e Antenne Médicale, Sarrebourg
  - Hôpital d'Instruction des Armées Sainte-Anne, Toulon
  - 60e Antenne Médicale, Valdahon

IPD SHARING:
Plan to Share IPD: Undecided